CLINICAL TRIAL: NCT05775991
Title: Enhancing Triadic Communication About Cognition for Older Adults With Alzheimer's Disease or Related Dementias Facing a Cancer Management Decision - Focus Groups
Brief Title: COACH-Cog Intervention Adaptation Focus Groups
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Allison Magnuson, Associate Professor of Medicine, University of Rochester
Other Study IDs: UOCPC22008; R01AG077053 (NIH)
Record Dates: First submitted 2023-01-20; First posted 2023-03-20 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Medical Oncologists and Clinicians: Individuals practicing as medical oncologists or with expertise in medical oncology. Clinicians with expertise in cognitive impairment and dementia
- Older patients with cancer: Older patients with cancer or older survivors of patients with cancer
- Caregivers of patients with dementia or cognitive impairment: Caregivers of patients with dementia or cognitive impairment

SUMMARY:
To gather key stakeholder input for feedback on the adaption of the COACH GA intervention (i.e., develop COACH-Cog) to enhance triadic communication among oncologists, care partners and patients with ADRD.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

The inclusion and exclusion criteria for participants are that they must be able to consent for themselves and must speak English.

For the medical oncologist focus group, participants must be a medical oncologist.

For the clinicians with expertise in cognitive impairment and dementia focus group, participants must be a clinician that treats patients with cognitive impairment and dementia.

For the older patients with cancer focus group, participants must be older than 65 years of age and have or had cancer.

For the caregivers of patients with dementia focus group, participants must be caregivers of patients with dementia or cognitive impairment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Focus groups will be conducted with the following stakeholders:
  1. Medical oncologists
  2. Clinicians with expertise in cognitive impairment and dementia
  3. Older patients with cancer
  4. Caregivers of patients with dementia
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Wilmot Cancer Institute, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Medical Oncologists and Clincians: Individuals practicing as medical oncologists or with expertise in medical oncology. Clinicians with expertise in cognitive impairment and dementia.
Period: Overall Study
Arm/Group | Medical Oncologists and Clincians | Older Patients With Cancer | Caregivers of Patients With Dementia or Cognitive Impairment
Started | 5 | 4 | 9
Completed | 5 | 4 | 7
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medical Oncologists and Clinicians | Older Patients With Cancer | Caregivers of Patients With Dementia or Cognitive Impairment | Total
Number analyzed (Participants) | 5 | 4 | 9 | 18
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years Between 18 and 65 years Between 18 and 65 years Between 18 and 65 years | 4 | 0 | 4 | 8
  >=65 years | 0 | 4 | 5 | 9
  Unknown/Missing | 1 | 0 | 0 | 1
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 3 | 2 | 6 | 11
  Male | 1 | 2 | 2 | 5
  Intersex | 0 | 0 | 0 | 0
  None of these describe me | 0 | 0 | 0 | 0
  Prefer not to answer | 0 | 0 | 1 | 1
  Missing | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 4 | 4 | 6 | 14
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 4 | 7 | 13
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Analysis of Focus Group Audio-recording Transcripts. Open Coding Using Content Analysis Framework Will be Utilized to Assess Positive Regard for the Intervention and Potential Intervention Adaptations.
Description: Qualitative data gathered from participants during focus group participation. Focus groups will be audio-recorded and transcribed. Transcribed audio-recordings will be qualitatively analyzed for positive regard for the intervention and opportunities and recommendations for further intervention adaptation. Open coding using content analysis framework will be utilized for qualitative analysis.
Time Frame: Through study completion approximately 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Oncologists and Clinicians | Older Patients With Cancer | Caregivers of Patients With Dementia or Cognitive Impairment
Number analyzed (Participants) | 5 | 4 | 9
Participants
  Positive Quote Given | 4 | 3 | 4
  Negative Quote Given | 0 | 0 | 0
  No Quote Given Applicable | 1 | 1 | 3
  Withdrew | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: We collected data on any adverse events that occur during the focus group that are attributable to the focus group which was 1 week in duration.
Arm/Group | Medical Oncologists and Clinicians | Older Patients With Cancer | Caregivers of Patients With Dementia or Cognitive Impairment
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/9
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT05775991/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT05775991/ICF_001.pdf